CLINICAL TRIAL: NCT06511401
Title: C-PAIN: Catalyzing Pharmacogenomic Analysis for Informing Pain Treatment
Brief Title: Informing Pain Treatment Using Pharmacogenomic Analysis
Acronym: C-PAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB24-0700; 1R01HG012273-01A1 (NIH)
Record Dates: First submitted 2024-07-05; First posted 2024-07-22 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Adult Patients Who Are Receiving Oncologic Care
Keywords: Pharmacogenomic; Opioids
MeSH Terms: interventions — Pharmacogenomic Testing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PGx Arm (Experimental): PGX information is provided to clinicals to inform opioid dosing and selection.
  Interventions: Other: Pharmacogenomic (PGx) results.
- Control Arm (No Intervention): No PGX information provided opioid dosing and selection is according to standard of care.

INTERVENTIONS:
Other: Pharmacogenomic (PGx) results. — These results are designed to provide specific dosing information based on the participant's unique genetics/genomics.
  Arms: PGx Arm

SUMMARY:
This is a randomized, prospective study to evaluate the effects of preemptive pharmacogenomic (PGx) testing on opioid dosing decisions/selections and pain score in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Persons receiving ongoing oncology care at the University of Chicago Medical Center for whom near-future pain opioid pain medication therapy is anticipated
* Subjects must be at least 18 years of age.

Exclusion Criteria:

* Subjects taking an opioid at the time of enrollment, or within the past 30 days
* Subjects who are currently undergoing palliative radiation
* Subjects who have undergone, or are being actively considered for, bone marrow, liver or kidney transplantation.
* Subjects with a history of or active blood cancer (e.g., leukemia).
* Chronic kidney disease, as defined by Glomerular filtration rate (GFR) < 30/mL/min/1.73m2, due to the risk of decreased drug excretion.
* Liver dysfunction, as defined by the following laboratory values, due to the risk of decreased drug metabolism: Total bilirubin greater than or equal to1.5 mg/dL, Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) greater than or equal to 2.5 X upper limit of normal*. (*Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) \ greater than or equal to 5 X upper limit of normal if hepatic metastases are present).
* Inability to understand and give informed consent to participate in the opinion of the investigator
* Subjects who are known to be pregnant at the time of enrollment
* Subjects who have previously or are currently enrolled in another institutional pharmacogenomic genotyping study, or are known to have previously undergone pharmacogenomic genotyping for the gene(s) of interest via another commercial or other means.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2028-01-07 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Pain control. | 45 days
  Measuring changes in composite pain intensity rating via the numeric rating scale:
  * Brief Pain Inventory-Short Form (BPI-SF)
  * Score range: 0 (no pain) to 10 (most pain)
  * Composite pain intensity score (mean of worst, least, average, and current pain)
  From baseline to day 45 in patients receiving an index opioid prescription for codeine, tramadol, or hydrocodone.

SECONDARY OUTCOMES:
Pain Medication Regimen Changes | 45 days
  Pain medication regimen changes will be assessed for patients who were taking an opioid metabolized primarily by CYP2D6. Pain medication regimen changes from baseline to day 45. The timing of subsequent changes in pain regimes after initial opioid selection will also be recorded.
Hospitalization or Emergency Visit for Pain Control | 45 days
  The rates of hospitalization and emergency room visits for pain are examined with the rates of increased utilization of health care resources, such as emergency department visits, hospitalizations, and pain consultations. Rates of hospitalization or emergency room visits from baseline to day 45.
Cumulative Morphine Equivalents Required | 45 days
  Cumulative Morphine Equivalents will be defined as total amount of opioids taken by a patient that is converted into its morphine equivalent. Dose and frequency of each opioid given during 45 days after its index prescription will be considered during calculation to give final values, which will be compared to Cumulative Morphine Equivalents for Control arms treated per standard of care.
Type of First Opioid Prescribed | From enrollment until study end (up to 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Peter H O'Donnell, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No